CLINICAL TRIAL: NCT02690519
Title: A Phase IIa, Open-label Study of Two Doses of GLPG1837 in Subjects With Cystic Fibrosis and the S1251N Mutation
Brief Title: Study of GLPG1837 in Subjects With Cystic Fibrosis (S1251N Mutation)
Acronym: SAPHIRA2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG1837-CL-202; 2015-003292-30 (EudraCT Number)
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis S1251N mutation; GLPG1837
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GLPG1837 dose 1 and GLPG1837 dose 2 (Experimental): GLPG1837 twice daily oral dosing - morning and evening, for 4 weeks
  Interventions: Drug: GLPG1837 dose 1; Drug: GLPG1837 dose 2

INTERVENTIONS:
Drug: GLPG1837 dose 1 — one GLPG1837 tablet in the morning and one GLPG1837 tablet in the evening, for 2 weeks
Drug: GLPG1837 dose 2 — one GLPG1837 tablet in the morning and one GLPG1837 tablet in the evening, for 2 weeks

SUMMARY:
At least 6 cystic fibrosis patients with the S1251N mutation will be treated for 4 weeks, consisting of two consecutive treatment periods of two weeks evaluating one dose of GLPG1837 each. After the treatment period, there is a 7-10 days follow-up period.

During the course of the study, subjects will be examined for any side effects that may occur (safety and tolerability).

Changes in sweat chloride will be assessed as biomarker from baseline onwards, and changes in pulmonary function (efficacy) will be explored throughout the study. The amount of GLPG1837 present in the blood (pharmacokinetics) will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age, with a confirmed diagnosis of cystic fibrosis
* Subjects with gating S1251N CFTR mutation on at least one allele in the CFTR gene
* Subjects currently receiving treatment with ivacaftor on a stable regimen or not on a treatment regimen with ivacaftor, for at least 2 weeks prior to screening
* Weight ≥ 40.0 kg
* Subjects on stable concomitant treatment regimen for at least 4 weeks prior to baseline (excluding ivacaftor)
* Pre- or post-bronchodilator FEV1 ≥ 40% of predicted normal
* Subject will have to use highly effective contraceptive methods

Exclusion Criteria:

* On an ivacaftor-containing treatment regimen and unable or unwilling to discontinue ivacaftor for the washout and treatment periods of the study
* Concomitant use of antifungal drugs within 4 weeks of baseline
* A history of a clinically meaningful unstable or uncontrolled chronic disease
* Liver cirrhosis and portal hypertension
* Any significant change in the medical regimen for pulmonary health within 4 weeks of baseline
* Unstable pulmonary status or respiratory tract infection or changes in therapy for pulmonary disease within 4 weeks of baseline
* Abnormal liver function
* Clinically significant abnormalities on ECG
* History of malignancy, solid organ/haematological transplantation
* Abnormal renal function
* Participation in another experimental therapy study within 30 days or 5 times half-life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes in adverse events | Up to 9 weeks
  To evaluate the safety and tolerability of GLPG1837 in terms of adverse events at every visit
Changes in laboratory parameters | Up to 7 weeks
  To evaluate the safety and tolerability of GLPG1837 in terms of abnormal laboratory parameters at every visit
Changes in vital signs | Up to 9 weeks
  To evaluate the safety and tolerability of GLPG1837 in terms of abnormal vital signs at every visit
Changes in physical examination | Up to 9 weeks
  To evaluate the safety and tolerability of GLPG1837 in terms of abnormal physical examination at every visit
Changes in electrocardiogram | Up to 7 weeks
  To evaluate the safety and tolerability of GLPG1837 in terms of abnormal electrocardiogram at every visit

SECONDARY OUTCOMES:
Changes in sweat chloride concentration | Up to 9 weeks
  To evaluate the effect of GLPG1837 in terms of change in sweat chloride concentration, a biomarker to measure cystic fibrosis transmembrane conductance regulator (CFTR) ion channel function at every visit
Changes in pulmonary function (forced expiratory volume in 1 second, FEV1) assessed by spirometry | Up to 9 weeks
  To explore the effect of GLPG1837 in terms of change in pulmonary function (forced expiratory volume in 1 second, FEV1) assessed by spirometry at every visit
Plasma levels of GLPG1837 | Up to 4 weeks
  To characterize the pharmacokinetics (PK) of GLPG1837 by measuring the amount in plasma between Day 1 and Day 29 at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Van de Steen, MD, MBA, Study Director — Galapagos NV
Locations (5):
- Belgium (3):
  - University Hospital Antwerp, Antwerp
  - University Hospital Ghent, Ghent
  - University Hospitals Leuven, Leuven
- Netherlands (2):
  - AMC, Amsterdam
  - UMC Utrecht, Utrecht